CLINICAL TRIAL: NCT01273662
Title: Axitinib as Second-line Treatment for Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Tri-Service General Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201008013M
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Axitinib (Experimental)
  Interventions: Drug: AG-013736

INTERVENTIONS:
Drug: AG-013736 — All enrolled patients will receive axitinib, 5 mg orally twice daily with food, until objective disease progression, development of unacceptable toxicity, or voluntary discontinuation by the subjects.
  Other Names: Axitinib

SUMMARY:
This is a phase II study of axitinib as the second-line on the treatment of advanced hepatocellular carcinoma (HCC).

The purpose of this study is a proof-of-concept study to see if axitinib has any anti-tumor effect in HCC. The primary endpoint is disease stabilization that lasts for at least 8 weeks without progression of tumor-related symptoms.

DETAILED DESCRIPTION:
Axitinib can can inhibit the activity of multiple angiogenesis-related signaling pathways. Promising anti-tumor activity has been demonstrated in patients with renal cell carcinoma, thyroid cancer, and melanoma. The potent anti-angiogenic activity of axitinib makes it a promising agent for the treatment of HCC.

This is a single-arm, open-label phase II trial. Eligible patients will receive axitinib, starting at 5 mg orally twice daily in the fasting status, until objective disease progression, development of unacceptable toxicity, or voluntary discontinuation. Dose titration will be done according to the severity of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed HCC, OR clinically diagnosed HCC
* Inoperable tumor(s) and no applicable curative therapy. Not amenable to loco-regional therapy
* Documented progression with or intolerance to sorafenib treatment as first- line therapy for advanced HCC
* At least one measurable tumor, according to RECIST version 1.1, that has not been treated with any local procedure
* ECOG performance status 0 or 1
* Life expectancy is at least 2 months
* Child-Pugh class A liver function.

Exclusion Criteria:

* Systemic therapy other than sorafenib as first-line therapy for advanced HCC
* History of HCC tumor rupture
* Presence of brain or leptomeningeal metastases
* Esophageal/gastric varices or active peptic ulcers that are considered to have high risk of bleeding
* History of upper gastrointestinal bleeding within 1 year
* Major systemic diseases that the investigator considers inappropriate for participation
* Uncontrollable hypertension
* Proteinuria
* Current use or anticipated need for treatment with potent CYP3A4 inhibitor, CYP3A4 or CYP1A2 inducers
* Requirement of anticoagulant therapy with oral vitamin K antagonists
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation and in the judgment of the investigator would make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
disease stabilization | 8 weeks until tumor progression

SECONDARY OUTCOMES:
time-to-tumor progression | 8 weeks until tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Lii Cheng, MD, PhD, Principal Investigator — Director/Professor
Locations (3):
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei